CLINICAL TRIAL: NCT03471988
Title: A Phase 3, Multi-center, Open Label Study to Evaluate Safety and Efficacy of AK1820 for Treatment of Adult Japanese Patients With Deep Mycosis
Brief Title: Clinical Study of AK1820 (Isavuconazonium Sulfate) for the Treatment of Deep Mycosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asahi Kasei Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK1820-301
Record Dates: First submitted 2018-02-26; First posted 2018-03-21 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-01

CONDITIONS: Deep Mycosis
Keywords: deep mycosis; aspergillosis; mucormycosis; cryptococcosis; isavuconazonium sulfate; isavuconazole; AK1820; Cresemba
MeSH Terms: conditions — Aspergillosis; Mucormycosis; Cryptococcosis | interventions — isavuconazole; Voriconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK1820 (Experimental): Participants will receive a loading dose of isavuconazole, 200 mg three times a day by intravenous infusion (IV) or orally for the first 2 days followed by a maintenance dose from Day 3 of 200 mg once daily either IV or orally until they will reach a treatment endpoint or for a maximum of 84 days.
  Interventions: Drug: AK1820
- Voriconazole (Active Comparator): Participants will receive a loading dose of voriconazole, 6 mg/kg every 12 hours IV or 300 mg every 12 hours orally for the first 24 hours, followed by a maintenance dose from Day 2 of 4 mg/kg every 12 hours by IV or 200 mg every 12 hours orally, until they will reach a treatment endpoint or for a maximum of 84 days.
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: AK1820 — Only a switch from IV infusion (vial) to oral administration (capsule) will be permitted; a switch from oral administration to IV infusion will not be possible.
  372.6 mg of AK1820 (isavuconazonium sulfate) is equivalent to 200 mg of isavuconazole.
  Other Names: Cresemba, BAL8557
  Arms: AK1820
Drug: Voriconazole — Only a switch from IV infusion (vial) to oral administration (tablet) will be permitted; a switch from oral administration to IV infusion will not be possible.
  Other Name : VFend
  Arms: Voriconazole

SUMMARY:
The objective of this study is to investigate the safety and efficacy of administering 372.6 mg of AK1820 (isavuconazonium sulfate) intravenously or orally to adult Japanese patients with deep mycosis. The primary endpoint is safety (percentage of patients with adverse events after starting the study treatment).

ELIGIBILITY:
Main Inclusion Criteria:

* Patients must have the below proven, probable or possible deep mycosis;

  1. invasive aspergillosis
  2. chronic pulmonary aspergillosis
  3. mucormycosis
  4. cryptococcosis
* Female patients must be non-lactating and at no risk for pregnancy.

Main Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Patients with hypersensitivity to any of the components of the azole class of antifungals or the investigational product.
* Patients at high risk for QT/QTc prolongation, or patients with risk factors for torsades de pointes, or taking concomitant medications known to prolong the QT/QTc interval.
* Patients with a history of short QT syndrome.
* Patients with liver dysfunction at enrollment.
* Patients with moderate to severe kidney dysfunction at enrollment.
* Patients who receive prohibited concomitant drugs.
* Patients with any other fungal infection other than Aspergillus species, order Mucorales, or Cryptococcus species.
* Patients who are not expected to survive study duration.
* Patients with an underlying disease, complication or general condition that would complicate safety and efficacy evaluations.
* Patients with a history of taking voriconazole for deep mycosis and showing no response to this treatment.
* Patients taking systemic antifungals who are unable to stop taking these drugs during the study, or who are showing signs of improvement in their symptoms of deep mycosis as a result of these drugs.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with adverse events between the first administration of investigational product and the end of Follow-up. | From the first study drug administration until 28 days after the last dose of study drug (up to approximately Day 112).

SECONDARY OUTCOMES:
Percentage of participants with an overall outcome of success evaluated by the data review committee (DRC). | Day 42, Day 84 and End of Treatment* (maximum Day 84).*End of treatment (EOT) is defined as the last day of study drug treatment.
Percentage of participants with clinical, radiological and mycological response assessed by the DRC. | Day 42, Day 84 and End of Treatment* (maximum Day 84).*End of treatment (EOT) is defined as the last day of study drug treatment.
Percentage of participants with overall outcome, clinical, radiological and mycological response evaluated by investigator. | Day 42, Day 84 and End of Treatment* (maximum Day 84).*End of treatment (EOT) is defined as the last day of study drug treatment.
All-cause mortality. | Through 28 days after the last dose of study drug (up to approximately Day 112).

CONTACTS AND LOCATIONS:
Locations (33):
- Japan (33):
  - Research site, Nagakute, Aichi-ken
  - Research site, Nagoya, Aichi-ken
  - Research site, Seto, Aichi-ken
  - Research site, Higashiku, Fukuoka
  - Research site, Minamiku, Fukuoka
  - Research site, Nagara, Gifu
  - Research site, Naka-Ku, Hiroshima
  - Research site, Asahikawa, Hokkaido
  - Research site, Kawasaki, Kanagawa
  - Research site, Yokohama, Kanagawa
  - Research site, Chuo-Ku, Kumamoto
  - Research site, Tsu, Mie-ken
  - Research site, Isahaya, Nagasaki
  - Research site, Ōmura, Nagasaki
  - Research site, Sasebo, Nagasaki
  - Research site, Tenri, Nara
  - Research site, Yufu, Oita Prefecture
  - Research site, Kurashiki, Okayama-ken
  - Research site, Nakagami, Okinawa
  - Research site, Abeno-Ku, Osaka
  - Research site, Sakai, Osaka
  - Research site, Ōmiya, Saitama
  - Research site, Hamamatsu, Shizuoka
  - Research site, Shimotsuke, Tochigi
  - Research site, Kiyose, Tokyo
  - Research site, Minato-Ku, Tokyo
  - Research site, Mitaka, Tokyo
  - Research site, Ōta-ku, Tokyo
  - Research site, Shinagawa-Ku, Tokyo
  - Research site, Shinjuku-Ku, Tokyo
  - Research site, Chiba
  - Research site, Ibaraki
  - Research site, Nagasaki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kohno S, Izumikawa K, Takazono T, Miyazaki T, Yoshida M, Kamei K, Ogawa K, Taniguchi S, Akashi K, Tateda K, Mukae H, Miyazaki Y, Okada F, Kanda Y, Kakeya H, Suzuki J, Kimura SI, Kishida M, Matsuda M, Niki Y. Efficacy and safety of isavuconazole against deep-seated mycoses: A phase 3, randomized, open-label study in Japan. J Infect Chemother. 2023 Feb;29(2):163-170. doi: 10.1016/j.jiac.2022.10.010. Epub 2022 Oct 25. PMID 36307059
- [Derived] Shirae S, Ose A, Kumagai Y. Pharmacokinetics, Safety, and Tolerability of Single and Multiple Doses of Isavuconazonium Sulfate in Healthy Adult Japanese Subjects. Clin Pharmacol Drug Dev. 2022 Jun;11(6):744-753. doi: 10.1002/cpdd.1079. Epub 2022 Feb 21. PMID 35191210